CLINICAL TRIAL: NCT03433443
Title: The Effect and Cost-effectiveness of a Case Manager to Assist the Rehabilitation of Lumbar Spinal Fusion Patients. A Randomised Controlled Trial.
Brief Title: Effect of a Case Manager to Assist the Rehabilitation for Lumbar Spinal Fusion Patients. A Randomised Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAarhus_CM_rehab
Record Dates: First submitted 2018-02-01; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Rehabilitation; Spinal Fusion; Case Managers
Keywords: Spinal Fusion; Case Managers; Rehabilitation

STUDY DESIGN:
Masking Description: Due to the nature of this study it was not possible to mask the participants, care providers or the investigator. We did not use any objective outcome measures assessed by outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Usual physical rehabilitation group
  Interventions: Behavioral: Usual physical rehabilitation
- Intervention group (Experimental): Case manager assisted rehabilitation
  Interventions: Behavioral: Case manager assisted rehabilitation; Behavioral: Usual physical rehabilitation

INTERVENTIONS:
Behavioral: Case manager assisted rehabilitation — In addition to receiving usual physical rehabilitation the patients in the intervention group had a case manager assigned. A team of three case managers delivered the intervention: a medical doctor specialized in social medicine, an occupational therapist, and a social worker. The case managers were all experienced case managers for non-surgical low back pain patients. The allocation to the case manager was random, and all patients had a main case manager assigned. The case managers involved the other case managers if their special knowledge were needed. Barriers for the patient's rehabilitation were discussed with the multidisciplinary team also including a surgeon, a physiotherapist, and a nurse.
  Arms: Intervention group
Behavioral: Usual physical rehabilitation — The patients received usual physical rehabilitation at their community rehabilitation unit, and had no case manager assigned.

SUMMARY:
The aim of the current study is to examine the effect of a case manager-assisting rehabilitation program compared to usual physical rehabilitation for patients undergoing a lumbar spinal fusion on functional disability, pain, and return to work. Furthermore, to explore if the case manager-assisted rehabilitation program is cost-effective in a societal perspective compared to usual rehabilitation.

Participants: 82 patients undergoing a lumbar spinal fusion due to disc degeneration or spondylolisthesis. Participants are adults of both gender.

Patients are included from Aarhus University Hospital, Denmark, and Region Hospital of Silkeborg, Denmark. Participants will be block randomised at each centre. The participants were randomized 1:1 to case manager-assisted rehabilitation (intervention group) or usual physical rehabilitation (control group). Both groups received usual physical rehabilitation. The patients in the intervention group meet pre-operatively with a case manager in order to set a plan for their return to daily activities and work. The intervention also included post-surgical meetings, phone meetings, work place visits, or voluntary roundtable meetings.

DETAILED DESCRIPTION:
The past decades have seen an increase in the numbers of patients undergoing lumbar spinal surgery due to degenerative diseases in the lumbar spine. The return to work rates following a lumbar spinal fusion have been reported to be between 35 and 50 percentages one year after the surgery and between 50-63% at 2-3-year after the surgery.

The aim of the current study is to examine the effect of a case manager-assisting rehabilitation program compared to usual physical rehabilitation for patients undergoing a lumbar spinal fusion on functional disability, pain, and return to work. Furthermore, to explore if the case manager-assisted rehabilitation program is cost-effective in a societal perspective compared to usual rehabilitation.

A total of 82 patients were included from Aarhus University Hospital, Denmark, and Region Hospital of Silkeborg, Denmark. Participants were block randomised at each centre. The participants were randomized 1:1 to case manager-assisted rehabilitation (intervention group) or usual physical rehabilitation (control group), by use of sealed envelopes. Both groups received usual physical rehabilitation. The patients in the intervention group meet pre-operatively with a case manager in order to set a plan for their return to daily activities and work. The intervention also included post-surgical meetings, phone meetings, work place visits, or voluntary roundtable meetings.

Statistical analysis:

For the power calculation, the Oswestry Disability Index was used. Based on another study in process at the time of the planning of the study, and in accordance to other research the standard deviation was set to 17 points. With a minimal clinical important difference of 12 points, a power of 80%, and a two sided significance level of 0.05, a total of 66 patients (33 in each group) should be included. I order to account for a 20% lost to follow-up a total om 80 patient should be included.

Data will be entered twice into EpiData and any divergence will be corrected according to the original material. STATA 14.1 will be used for statistical evaluation. The risk of a type 1 error was set to 5%. The data will be analyzed according to the intention-to-treat principle.

I order to compare the two groups a mixed model for repeated measurements with an unstructured covariance matrix will be used to test the effect on Oswestry Disability Index, back pain, and leg pain.

I order to evaluate the patients' return to work following the surgery, the cumulative incidence proportion of time to first spell of 4 weeks of return to work within a 2-year period will be calculated and compared by the log rank test. The relative cumulative incidens of a spell of 4 weeks' return to work will be analysed in a generalized linear regression model using the pseudo values method adjusted for time until old age pension and disability pension.

The primary outcome used in the economic evaluation are functional disability as measured by the Oswestry Disability Index. Furthermore, health-related quality of life was measured by the EuroQol 5-dimensions (EQ-5D) and valued by Danish preference weights in order to calculate Quality Adjusted Life Years (QALY).

The resource use, costs, and outcomes will be analysed as arithmetic means with 95% bootstrapped confidence intervals based on non-parametric bootstrapping (10,000 replicates), and after discounting at an annual rate of 3%. To assess the cost-effectiveness, costs and outcomes will be transformed into a uni-dimensional measure of incremental net benefit for a range of hypothetical values of willingness to pay per unit of effect: incremental net benefit = (EA - EB) * willingness to pay per effect unit - (CA - CB), where C denotes costs and E denotes effects with A and B referring to comparators.

The study protocol was approved by the Danish Data Protection Agency (J.nr.2010-41-444), and the local Ethical Committee (J.nr.M-20100038)

ELIGIBILITY:
Inclusion Criteria:

* All patients were scheduled for an lumbar spinal fusion due to degenerative disc disease or spondylolisthesis grade I or II.

Exclusion Criteria:

* age below 18 years or above 63 years, inability to speak and understand Danish, a driving distance of more than 100 kilometers to the hospital, un-instrumented lumbar spinal fusion, disability pension, early retirement, being out of the working force for more than 24 months, and patients under education on State education grant.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2011-10-01 (Actual); Study Completion 2014-11-05 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (functional disability) | The time frame was two years (measured from baseline to two years follow-up). Intermediate follow-up at three months, six months, nine months, one year after surgery.
  Patient reported questionnaire to measure functional disability. Scoring from 0 - 100, 0=no problems, 100=most problems. We will compare changes from baseline to two year follow-up between the two groups.

SECONDARY OUTCOMES:
Low Back Pain Rating Scale (measuring back and leg pain) | The time frame was two years (measured from baseline to two years follow-up). Intermediate follow-up at three months, six months, nine months, one year after surgery.
  Patient reported questionnaire to measure back pain and leg pain on two separated sub-scales one for back pain and one for leg pain. The sub-scales ranges from 0-10, 0=no pain, 10=worst pain. We will compare changes from baseline to two year follow-up between the two groups.
Return to work rates | The time frame was two years (measured from baseline to two years follow-up)
  Use of the national register the Danish Register for Evaluation of Marginalization (DREAM) in order to measure the cumulative incidence proportion of time to first spell of four weeks of return to work within a two-years period. The register list employment status for each week on an individual level. We will compare changes from baseline to two year follow-up between the two groups.
EuroQol 5-dimensions (Quality of Life) | The time frame was two years (measured from baseline to two years follow-up). Intermediate follow-up at three months, six months, nine months, one year after surgery.
  The EuroQol 5-dimensions will be valued by Danish preference weights. Patient reported questionnaire to measure quality of life on a scale from -0.56 - 1.0. -0.56=worst possible health. 1.0 = health as a new-born. The EuroQol 5-dimensions scores will be used to calculate the Quality Adjusted Life Years as the areas under the curve. We will compare changes from baseline to two year follow-up between the two groups.
Number of weeks on sick leave | The time frame was two years (measured from baseline to two years follow-up)
  Use of the national register the Danish Register for Evaluation of Marginalization (DREAM) in order to measure number of weeks of sick leave within a two-years period. The register list employment status for each week on an individual level. We will compare numbers of weeks of sick leave between the two groups.

OTHER OUTCOMES:
Number of hours of help in the home | The time frame was one year (measured from baseline to one year follow-up)
  Questionnaire to measure the patient reported use of health care services including help from family and friend, private home care, private domestic help. The measures is numbers of hours. The outcome measure will be use in the planned economic evaluation.
Numbers of hospital out patients visits | The time frame was two years (measured from baseline to two years follow-up)
  Numbers of contacts extracted from the National Patient Registry. The outcome measure will be use in the planned economic evaluation.
Numbers of contacts to private physiotherapists | The time frame was two years (measured from baseline to two years follow-up)
  Numbers of contacts extracted from The National Health Insurance Service Register. The outcome measure will be use in the planned economic evaluation.
Number of contacts to medical specialist in primary care | The time frame was two years (measured from baseline to two years follow-up)
  Numbers of contacts extracted from The National Health Insurance Service Register. The outcome measure will be use in the planned economic evaluation.
Number of contacts to general practitioner | The time frame was two years (measured from baseline to two years follow-up)
  Numbers of contacts extracted from The National Health Insurance Service Register. The outcome measure will be use in the planned economic evaluation.
Number of days admitted to hospital | The time frame was two years (measured from baseline to two years follow-up)
  Numbers of days extracted from the National Patient Registry. The outcome measure will be use in the planned economic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa G Østergaard, Principal Investigator — Aarhus University Hospital, Department of Physiotherapy and Occupational Therapy

IPD SHARING:
Plan to Share IPD: No
Only individual participant data that are made available in published papers.